CLINICAL TRIAL: NCT06545903
Title: Supraglottic Airway Devices for Airway Management of Entrapped Trauma Patients - an Evaluation of Four Devices in a Simulated Condition With Simultaneous Cervical Spine Immobilisation - a Randomised, Controlled Trial
Brief Title: Supraglottic Airways for Entrapped Trauma Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Uniwersytet Radomski im. Kazimierza Pułaskiego (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: 3/2024
Record Dates: First submitted 2024-07-16; First posted 2024-08-09 (Actual); Last update posted 2025-05-06 (Actual); Status verified 2025-05

CONDITIONS: Airway Obstruction
Keywords: Entrapped Trauma Patients; Airway Management; Paramedics
MeSH Terms: conditions — Airway Obstruction

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- LMA Supreme Group (Active Comparator): Paramedics using the LMA Supreme airway device
  Interventions: Device: LMA Supreme
- Other Supraglottic Airway Group (Experimental): Paramedics using other supraglottic devices
  Interventions: Device: SLIPA; Device: I-gel; Device: AuraGain

INTERVENTIONS:
Device: LMA Supreme — The device is inserted and the manikin ventilated
  Arms: LMA Supreme Group
Device: SLIPA — The device is inserted and the manikin ventilated
  Arms: Other Supraglottic Airway Group
Device: I-gel — The device is inserted and the manikin ventilated
  Arms: Other Supraglottic Airway Group
Device: AuraGain — The device is inserted and the manikin ventilated
  Arms: Other Supraglottic Airway Group

SUMMARY:
The aim of this clinical trial is to evaluate four supraglottic airway devices for ventilation in a simulated condition of an entrapped trauma patient with simultaneous cervical spine immobilisation. All the studied devices are evaluated by fully-qualified and experienced paramedics (both male and female). The main questions it aims to answer are:

1. Which device requires the shortest time required to achieve a successful ventilation?
2. What is the first attempt success rate of the studied devices?
3. Which device is the easiest to use and the most user-friendly? Study participants will evaluate four different supraglottic devices in a restricted access to the entrapped trauma patient's airway. The maximum number of insertion attempts is limited to three per device.

DETAILED DESCRIPTION:
A 10-minute lecture will be delivered before the start of the study. It will explain how to use the studied devices. Following the lecture all participants will be able to familiarise themselves with the equipment and practice for 30 minutes. A skill station will be set up containing an intubation manikin AT Kelly Torso (Laerdal Medical AS, Stavanger, Norway). A reduced movement of the cervical spine will be achieved by application of a Patriot® cervical collar (Össur hf., Reykjavik, Iceland). After completion of the initial practice the intubation manikin with the cervical collar on will be placed on and secured to the driver's seat of a medium-sized passenger car (FIAT S.p.A., Turin, Italy). The car will then be positioned on its left side and secured in place by firemen from a local fire brigade. The access to the manikin will only be allowed from the front i.e. through the opening created after removal of the windscreen. A single digit number will be allocated to each of the four studied devices i.e. 1 for the SLIPA device, 2 for the I-gel, 3 for the LMA Supreme and 4 for the LTS. Each study participant will be asked to randomly give a number (either 1, 2, 3 or 4) and will then be given the corresponding airway device to use. The maximum number of insertion attempts will be limited to three per device. The time required to insert the device and achieve a successful ventilation (Tiv) will be recorded. It will be measured using a stopwatch of a mobile phone (Apple Inc., Cupertino, California, USA). Efficacy of insertion/ventilation and the ease of use by the operator will also be assessed. The latter will be measured using an 11-point numerical rating scale (NRS) where 0 corresponds to a very difficult to use device and 10 indicates an easy to use and user-friendly device. A manual resuscitator (Ambu A/S, Ballerup, Denmark) will be used for ventilation and will be readily available to the paramedics. The study participants will perform all insertions with each of the four supraglottic airway devices. A failed insertion and ventilation is defined as an attempt during which the manikin cannot be ventilated or an attempt that lasted longer than 120 seconds. Only those who failed to ventilate will be allowed another attempt. All the obtained data will be analysed using Microsoft Office Excel 2021 spreadsheet (Microsoft Corporation, Redmond, WA, USA). The Kolmogorov-Smirnov test is utilised to determine whether the analysed variables matched the characteristics of a normal distribution. A paired Student t-test and the Wilcoxon signed-rank test will be used for data analysis. Based on our previous unpublished pilot study and assuming that the overall success rate of intubation in patients with a difficult airway would be 90% (α =0.05, 2-sided, β =0.1), 46 participants will be required. The final adjusted sample size, allowing a drop-out rate of about 10%, is 50 and this is the final number of participants enrolled into the study. A p-value of less than 0.05 (p<0.05) is considered statistically significant.

ELIGIBILITY:
Inclusion Criteria:

* fully-qualified paramedics
* at least four years of practice after finishing paramedic training
* active (working) paramedics

Exclusion Criteria:

* paramedics in training
* retired paramedics
* lack of written informed consent

Ages: 25 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 50 (Actual)
Dates: Start 2024-07-01 (Actual); Primary Completion 2024-09-01 (Actual); Study Completion 2025-05-01 (Actual)

PRIMARY OUTCOMES:
Successful ventilation time | During procedure: 120 seconds
  The time required to insert the device and achieve a successful ventilation

SECONDARY OUTCOMES:
First attempt success rate of ventilation | During procedure: 120 seconds
  The efficacy of an evaluated supraglottic airway device
The ease of use and user-friendliness | During procedure: 120 seconds
  Device evaluation using the numerical rating scale (NRS). It is an 11-point scale where 0 corresponded to a very difficult to use device and 10 indicated an easy to use and user-friendly device.

CONTACTS AND LOCATIONS:
Overall Officials: Dawid J Aleksandrowicz, PhD, Principal Investigator — University of Radom
Locations (1):
- University of Radom, Radom, Masovian Voivodeship, Poland

IPD SHARING:
Plan to Share IPD: No